CLINICAL TRIAL: NCT00940017
Title: A Phase 4, Open Label Study To Assess The Bronchopulmonary Pharmacokinetics Of Anidulafungin And Voriconazole Following Intravenous Administration In Healthy Subjects
Brief Title: A Study To Assess The Anidulafungin And Voriconazole Concentration In Lung Following Intravenous Administration In Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: A8851020
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-01

CONDITIONS: Aspergillosis; Candidemia
Keywords: PK; fungal infection
MeSH Terms: conditions — Aspergillosis; Candidemia; Mycoses | interventions — Anidulafungin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: anidulafungin and voriconazole

INTERVENTIONS:
Drug: anidulafungin and voriconazole — Subjects will be admitted to the clinical research unit on Day 0. Subjects will receive anidulafungin intravenously in a loading dose of 200 mg on Day 1, followed by maintenance doses of 100 mg Q24h on Day 2 and Day 3. Simultaneously, using a separate intravenous access, subjects will receive voriconazole in a loading dose of 6 mg/kg Q12h on Day 1, followed by a maintenance dose of 4 mg/kg Q12h on Day 2, and a 4 mg/kg morning dose on Day 3.

SUMMARY:
The purpose of this study is to provide anidulafungin and voriconazole to healthy subjects to determine the drug concentration in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects willing to comply with the study requirement.

Exclusion Criteria:

* Clinical significant disease.
* Sensitive to study medication.
* Not willing to comply with the study requirement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hartford, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851020&StudyName=A%20Study%20To%20Assess%20The%20Anidulafungin%20And%20Voriconazole%20Concentration%20In%20Lung%20Following%20Intravenous%20Administration%20In%20Healthy%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin and Voriconazole: Anidulafungin (Eraxis™) intravenously (IV) in a loading dose of 200 milligrams (mg) on Day 1, followed by maintenance doses of 100 mg every 24 hours on Day 2 and Day 3. Simultaneously, using a separate intravenous access, subjects received voriconazole (Vfend®) in a loading dose of 6 milligrams per kilogram (mg/kg) every 12 hours on Day 1, followed by a maintenance dose of 4 mg/kg every 12 hours on Day 2, and a 4 mg/kg morning dose on Day 3.
Period: Overall Study
Arm/Group | Anidulafungin and Voriconazole
Started | 24
Subjects Treated | 21
Completed | 20
Not Completed | 4
Not completed — did not meet entrance criteria | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax)
Description: Cmax = maximum observed plasma concentration; measured in micrograms per milliliter (ug/mL). Observed directly from the data. Collected on Day 3.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
ug/mL
  Anidulafungin | 6.56 (1.62)
  Voriconazole | 5.32 (1.82)

2. Primary Outcome: Plasma PK: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax = time (hours) to maximum plasma concentration (Cmax). Observed directly from data as time of first occurrence. Collected on Day 3.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population
Measure: Median (Full Range); unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
hours
  Anidulafungin | 1.93 [1.70 to 2.17]
  Voriconazole | 1.74 [1.67 to 2.05]

3. Primary Outcome: Plasma PK: Area Under the Curve From Time Zero to Time = Tau (AUCtau)
Description: AUCtau = area under the plasma concentration-time profile from time zero (0) to time = t (AUCt), the dosing interval, where t is 24 hours for anidulafungin and 12 hours for voriconazole; measured as micrograms times hours per milliliter (ug*hr/mL). Collected on Day 3.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population defined as all subjects randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
ug*hr/mL
  Anidulafungin | 101 (21.8)
  Voriconazole | 39.5 (19.8)

4. Primary Outcome: Plasma PK: Plasma Elimination Half-life (t1/2)
Description: t1/2 = terminal elimination half-life in hours; Loge(2)/Kel, where Kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Collected on Day 3.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; (n) = number of subjects contributing to the mean
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 18
hours
  Anidulafungin (n=18) | 20.8 (3.06)
  Voriconazole (n=15) | 6.94 (2.10)

5. Primary Outcome: Plasma PK: Total Clearance (CL Total)
Description: CL total = total clearance calculated as dose divided by AUCt; measured as milliliters per minute (mL/min). Collected on Day 3.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
mL/min
  Anidulafungin | 17.1 (3.04)
  Voriconazole | 172 (86.2)

6. Primary Outcome: Plasma PK: Volume of Distribution at Steady-state (Vss)
Description: Vss = volume of distribution at steady-state; measured as liters (L). Calculated as (CL multiplied by mean residence time extrapolated to infinity [MRTinf]). MRTinf = [(AUMCt plus t (AUCinf minus AUCt)) divided by AUCt] minus (infusion time divided by 2); AUMCt = area under the first moment curve from time zero to time t; AUCinf = area under the plasma concentration-time curve extrapolated to infinity.
Time Frame: 100 minutes (end of infusion), 2, 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; (n) = number of subjects contributing to the mean.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 18
L
  Anidulafungin (n=18) | 30.8 (6.84)
  Voriconazole (n=15) | 110 (34.0)

7. Primary Outcome: Epithelial Lining Fluid (ELF) PK: Cmax
Description: Cmax=maximum observed plasma concentration. ELF collected by bronchoscopy and bronchoalveolar lavage (BAL) Day 3; determined from BAL sample using urea dilution method: [Drug ELF]=[Drug BAL] multiplied by [Urea SERUM] divided by [Urea BAL]. Drug ELF=anidulafungin or voriconazole (drug) concentration in ELF corrected for dilution; Drug BAL=assayed drug concentration in BAL; Urea SERUM and Urea BAL simultaneously collected. Summary parameters derived using average data for all subjects; associated to a single subject for reporting purposes (mean with standard deviation not calculated).
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: average concentration (ug/mL)
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
average concentration (ug/mL)
  Anidulafungin | 1.13
  Voriconazole | 48.3

8. Primary Outcome: ELF PK: Tmax
Description: Tmax = time (hours) to maximum plasma concentration (Cmax). Observed directly from data as time of first occurrence. ELF collected by bronchoscopy and BAL on Day 3.
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
hours
  Anidulafungin | 24.0
  Voriconazole | 4.0

9. Primary Outcome: ELF PK: AUCtau
Description: AUCtau = area under the plasma concentration-time profile from time zero (0) to time = t (AUCt), the dosing interval, where t is 24 hours for anidulafungin and 12 hours for voriconazole. ELF collected by bronchoscopy and BAL on Day 3. Summary parameters were derived using average data for all subjects and associated to a single subject for reporting purposes (mean with standard deviation was not calculated).
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: average concentration (ug*hr/mL)
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
average concentration (ug*hr/mL)
  Anidulafungin | 21.9
  Voriconazole | 282

10. Primary Outcome: ELF PK: t1/2
Description: t1/2 = terminal elimination half-life in hours; Loge(2)/Kel, where Kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. ELF collected by bronchoscopy and BAL on Day 3.
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects. Data in ELF did not allow calculation of t1/2; not analyzed.
Measure: Number; unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 0

11. Primary Outcome: Alveolar Macrophages (AM): Cmax
Description: Cmax = maximum observed plasma concentration; observed directly from the data. AM collected by bronchoscopy and BAL on Day 3. Summary parameters were derived using average data for all subjects and associated to a single subject for reporting purposes (mean with standard deviation was not calculated).
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: average concentration (ug/mL)
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
average concentration (ug/mL)
  Anidulafungin | 103
  Voriconazole | 20.5

12. Primary Outcome: AM: Tmax
Description: Tmax = time (hours) to maximum plasma concentration (Cmax). Observed directly from data as time of first occurrence. AM collected by bronchoscopy and BAL on Day 3.
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
hours
  Anidulafungin | 24
  Voriconazole | 4.0

13. Primary Outcome: AM: AUCtau
Description: AUCtau = area under the plasma concentration-time profile from time zero (0) to time = t (AUCt), the dosing interval, where t is 24 hours for anidulafungin and 12 hours for voriconazole. AM collected by bronchoscopy and BAL on Day 3. Summary parameters were derived using average data for all subjects and associated to a single subject for reporting purposes (mean with standard deviation was not calculated).
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: average concentration (ug*hr/mL)
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
average concentration (ug*hr/mL)
  Anidulafungin | 1430
  Voriconazole | 178

14. Primary Outcome: AM: t1/2
Description: t1/2 = terminal elimination half-life in hours; Loge(2)Kel, where Kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AM collected by bronchoscopy and BAL on Day 3.
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects. Data in AM did not allow calculation of t1/2; not analyzed.
Measure: Number; unit: hours
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 0

15. Primary Outcome: Overall Drug Penetration Ratio in ELF
Description: ELF collected by bronchoscopy and BAL on Day 3. ELF to plasma penetration ratio calculated by dividing area under the plasma concentration-time profile (AUC) in ELF by AUC in plasma from 20 subjects where t is 24 hours for anidulafungin and 12 hours for voriconazole. Summary parameters were derived using average data for all subjects and associated to a single subject for reporting purposes (mean with standard deviation was not calculated).
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects.
Measure: Number; unit: average ELF to plasma ratio
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
average ELF to plasma ratio
  Anidulafungin | 0.22
  Voriconazole | 7.14

16. Primary Outcome: Concentration Ratio in ELF to Plasma
Description: Concentration ratio in ELF to plasma determined by a point estimate within each subject at the time-point where ELF data was available.
Time Frame: 4, 8, 12, 24 hours after start of infusion
Population: PK parameter analysis population; summary parameters derived using average data for all subjects. Subjects randomized to a single BAL procedure timepoint; bronchoscopy and BAL done for 5 different subjects at each timepoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Anidulafungin and Voriconazole
Number analyzed (Participants) | 20
ratio
  Anidulafungin 4 hours | 0.15 (0.02)
  Anidulafungin 8 hours | 0.15 (0.07)
  Anidulafungin 12 hours | 0.20 (0.09)
  Anidulafungin 24 hours | 0.38 (0.14)
  Voriconazole 4 hours | 9.50 (2.31)
  Voriconazole 8 hours | 4.93 (2.79)
  Voriconazole 12 hours | 7.68 (3.41)

ADVERSE EVENTS:
Arm/Group | Anidulafungin and Voriconazole
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 15/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin and Voriconazole (N=21)
Photophobia (Eye disorders) | 2
Visual impairment (Eye disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Influenza like illness (General disorders) | 4
Hypersensitivity (Immune system disorders) | 1
Liver function test abnormal (Investigations) | 1
Headache (Nervous system disorders) | 6
Hallucination, visual (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.